CLINICAL TRIAL: NCT03771885
Title: A Phase Ib, Multicentre, Randomised, Double-blind, Placebo Controlled, 8 Week Crossover Study to Assess the Safety, Tolerability and Pharmacokinetics of Orally Administered BI 705564 in Patients With Systemic Lupus Erythematosus.
Brief Title: BI 705564 in Patients With Systemic Lupus Erythematosus (SLE)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Based on a strategic decision, the application for the trial has been withdrawn before initiation.
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1408-0004; 2017-004948-38 (EudraCT Number)
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Lupus Erythematosus, Systemic
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): 4 weeks place followed by 4 weeks IMP
  Interventions: Drug: BI 705564; Drug: Placebo
- Group B (Experimental): 4 weeks IMP followed by 4 weeks placebo
  Interventions: Drug: BI 705564; Drug: Placebo

INTERVENTIONS:
Drug: BI 705564 — Film-coated Tablet
Drug: Placebo — Film-coated Tablet

SUMMARY:
The main objective of this study is to assess the safety, tolerability and pharmacokinetics of orally administered BI 705564 in patients with systemic lupus erythematosus

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years at screening.
* Diagnosis of systemic lupus erythematosus (SLE) at least 6 months prior to screening according to SLICC 2012 criteria; at least 4 criteria must be documented.
* Positive test results for anti-nuclear antibody (ANA) (human epithelial cell-2 ANA greater than or equal to [>=] 1:80) and/or anti-dsDNA antibody at the Screening visit. To be performed by Central Laboratory.
* At screening visit a "clinical" Systemic Lupus Erythematosus Disease Activity Index (2K), (SLEDAI 2K) score of ≥ 4 points. The "clinical" score is the SLEDAI 2K assessment score without the inclusion of points attributable to any blood laboratory results including immunologic measures. Neurologic descriptors of the SLEDAI 2K are not counted towards the SLEDAI 2K study entry criteria.
* Has received all scheduled vaccines according to local guidelines and Investigator judgement. Live or live-attenuated virus vaccines are not permitted within 1 month prior to screening or during screening. For all other vaccines there must be at least 2 weeks between the vaccination(s) and the date of randomization at Day 1.
* For male patients: Men who are permanently sterile by bilateral orchidectomy are not required to use contraception. Men whose partner (or potential partner) is a women of childbearing potential*, for the duration of the study (including 30 days after the last dose of study drug) must use a condom. For female patients: Women of childbearing potential* must be willing and able to use a double-barrier contraception (barrier in the meaning of method) with at least one highly effective method of birth control per ICH M3(R2) that result in a low failure rate of less than 1% per year when used consistently and correctly for the duration of the study including 4 weeks after the last dose of study drug. Medically accepted methods of contraception in this study are:

  * Combined (oestrogen and progestogen containing) hormonal birth control associated with inhibition of ovulation in combination with male condom.
  * Progestogen-only hormonal birth control associated with inhibition of ovulation in combination with male condom.
  * Intrauterine device (IUD) and intrauterine hormone-releasing system (IUS) in combination with male condom Or

    * The patient must have only vasectomized sexual partner(s) (vasectomy at least 1 year prior to enrolment), Or
    * The patient must follow true abstinence from male-female sex. This is defined as being in line with the preferred and usual lifestyle of the patient. Periodic abstinence e.g. calendar, ovulation, symptothermal, post-ovulation methods; declaration of abstinence for the duration of exposure to IMP; and withdrawal are not acceptable.

      * A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. Tubal ligation is NOT a method of permanent sterilisation. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion Criteria:

* Active clinically significant neuropsychiatric SLE or any BILAG A score for a neuropsychiatric manifestation or in the ophthalmic domain within the past 12 months.
* Drug-induced Lupus.
* Other autoimmune diseases such as Rheumatoid Arthritis, Crohn's, scleroderma, psoriasis, Celiac disease, Graves'disease, thyroid disease, with the following exceptions:

  * Sjögren syndrome if this is secondary to their SLE is permissible.
  * Patients with features of mixed connective tissue disease may be included if this is secondary to their SLE and is, in the Investigator's opinion not considered to be significant.
  * Patients with APS antibodies may be included unless they are excluded due to exclusion anti-coagulation medication (see exclusion criteria below for details) or if they have a history of thromboembolic events or miscarriage.
  * Diabetes if this is considered by the Investigator to be well controlled and there is no evidence of retinopathy or nephropathy.
* Initiation or change in dose of anti-malarial treatment after the screening visit.
* Patients who require fibrinolysis, full-dose therapeutic anticoagulation (e.g. vitamin K antagonists, dabigatran, heparin, hirudin, etc.) or high dose antiplatelet therapy.
* Within 2 weeks prior to Screening or during Screening: use of oral corticosteroids greater than (>) 15 mg daily prednisone or an equivalent dose, use of any injectable corticosteroids, or change in dose of corticosteroids. For patients continuing on oral corticosteroids the dose must be stable for 4 weeks prior to randomisation.
* After consent, initiation or change in dose of angiotensin-converting enzyme inhibitor or angiotensin receptor blocker.
* Initiation of regular nonsteroidal anti-inflammatory drugs (NSAIDs) use within 2 weeks prior to Screening. Regular use defined as 3 consecutive days.
* Within 2 months prior to Screening or during Screening: initiation of or change in dose of methotrexate, mycophenolate (mofetil or sodium), or azathioprine.
* Within 4 weeks prior to Screening or during Screening, use of cyclosporine or tacrolimus.
* Within 3 months prior to Screening or during Screening: use of cyclophosphamide or chlorambucil.
* Within 3 months prior to Screening or during Screening, use of leflunomide, abatacept, anti-tumor necrosis factor alpha agents, intravenous immunoglobulin, plasmapheresis, or other disease modifying, immunosuppressive, or immunomodulatory therapies not otherwise specified in protocol.
* Within 12 months prior to screening or during screening: use of anti-CD20 or anti-CD22 biological medications or any other B cell-depleting medication. If a patient has had rituximab more than 6 months ago and has a normal CD-19 count then they may be included. A historic local lab value may be used to confirm this. For B-cell modulating therapies including atacicept these are excluded within 6 months apart from blisibimod and belimumab which are excluded within 3 months. Type I-IFN interferon antagonists such as anifrolumab are excluded within 6 months.
* Ustekinumab within 6 months of screening.
* JAK inhibitors within the last 12 months before screening visit.
* Active clinically significant viral, bacterial or fungal infection, or any serious episode of infection requiring hospitalization within the last 6 months. If the infection is not active or clinical significant or required hospitalization the patient may be included as long as they have not taken antibiotics more than 4 weeks prior to screening.
* Chronic Hepatitis B, HIV, history of active TB.

  * A patient with an indeterminate or positive TB test result at screening may be enrolled if a thorough investigation by a qualified physician determines that they do not have active TB or untreated latent TB.
  * In the case of Anti-HBc antibody positive result but HBs antigen negative then Hepatitis B DNA can be measured at a local lab. If Hepatitis B DNA is positive the patient will be excluded, if Hepatitis B DNA is negative then the patient can be included.
* Immunoglobulin G (IgG) less than the lower limit of normal at screening.
* Estimated glomerular filtration rate of less than (<) 60 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2) by the CKD-EPI (2009) Creatinine Equation, or recent decline in kidney function, defined as decrease within the last 2 months prior to screening:

  -- as a reduction in eGFR of >=20% and below lower limit of normal (90 mL/ min/ 1.73m2).
* Proteinuria > 2 g/d or urine protein/urine creatinine ratio >2 mg/mg at screening.
* Clinically significant other renal disease based on investigator judgement (e.g. postinfectious GN, pyelonephritis)
* Major surgery (major according to the investigator's assessment) performed within 12 weeks prior to randomization or planned during the trial.
* Any documented active or suspected malignancy or history of malignancy within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin or in situ carcinoma of uterine cervix.
* Patients who must or wish to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Previous randomisation into this trial.
* Currently enrolled in another investigational device or drug trial,

  * or less than 30 days or 5 half-lives (whichever is longer),since ending another investigational device or drug trial(s) for an oral agent which is not specified in any other exclusion criteria,
  * or less than 12 months since ending another investigational device or drug trial(s) for a biological agent which is not specified in exclusion criteria
  * or receiving other investigational treatment(s).
* Chronic alcohol or drug abuse or any condition that, in the investigator's opinion, makes them an unreliable trial patient or unlikely to complete the trial.
* Women who are pregnant, nursing, or who plan to become pregnant in the timeline of the trial.
* Uncontrolled hypertension or other haematologic conditions (except SLE). Diabetes mellitus if poorly controlled according to investigator or known diabetic nephropathy or retinopathy.
* Thrombocyte count at screening 70,000/μl or less.
* Known hypersensitivity to the study drug or their excipients.
* Patients with known ocular complications apart from dry eyes and mild cataracts in the opinion of an ophthalmologist.
* A disease or condition which in the opinion of the investigator may interfere with testing procedures or put the patient at risk when participating in this trial.
* History of pancreatitis of any aetiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-16 (Estimated); Primary Completion 2019-12-21 (Estimated); Study Completion 2020-01-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint to assess safety and tolerability of BI 705564 is the number of patients with drug related Adverse Events | Up to 73 Days

SECONDARY OUTCOMES:
Number and severity of Adverse Events | Up to 87 Days
Number of patients with Adverse Events | Up to 87 Days
Number of patients with Serious Adverse Events | Up to 87 Days
Change from baseline in BILAG | Up to 87 Days
Change from baseline in SLEDAI-2K | Up to 87 Days

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing